CLINICAL TRIAL: NCT03652987
Title: Evaluation of Endocrine and Menstrual Disturbances in Women With Polycystic Ovary Syndrome (PCOS): Impact of Weight, Metabolic Status, Age and Ethnicity.
Brief Title: Endocrine and Menstrual Disturbances in Women With Polycystic Ovary Syndrome (PCOS)
Acronym: EMDPCOS
Status: Suspended | Type: Observational
Why Stopped: Covid19-related restrictions
Sponsor: St George's, University of London (Other)
Collaborators: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: 18.0049
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2020-06

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance; Vitamin D Deficiency; Obesity
Keywords: PCOS; Hyperandrogenemia; Rotterdam Criteria; Insulin sensitivity; BMI; Antral follicle count
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Vitamin D Deficiency; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Urine and serum sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common endocrine disorder in reproductive age women, which causes disordered follicle growth and ovulation resulting in infertility. In addition women with PCOS have hyperandrogenemia and a dysregulated hormonal profile, resulting in altered feedback on the hypothalamic-pituitary-gonadal (HPG) axis. Obesity, insulin resistance, vitamin D (VD) deficiency and ageing worsen the symptoms. The gonadotrophins - follicle stimulating hormone (FSH) & luteinising hormone (LH), along with the pregnancy hormone human chorionic gonadotrophin (hCG) have structural similarities. The altered levels of FSH and LH in women with PCOS cause production of hCG from the brain leading to false positive pregnancy tests. Part one of this project will involve the investigation of this over-production of hCG in urine and serum of women with PCOS to develop suitable ovulation and pregnancy test kits, in collaboration with Swiss Precision Diagnostics (SPD). In Part two of the project, we would like to see if intervention with VD supplementation and/or using myo-inositol supplement compared with metformin (insulin sensitiser), improves prediabetes, distribution of fat/water content, weight loss and menstrual cyclicity in women with PCOS. We aim to correlate these interventions with particular serum & urine markers to develop better diagnostic tools.

DETAILED DESCRIPTION:
Women are referred by the general practioner (GP)/primary care with a suspected diagnosis of PCOS to the Endocrine Clinic at St George's Hospital.

They have an initial routine clinical assessment involving history, BP, weight & assessment of PCOS using the Rotterdam criteria.

The routine clinical investigations involve the following:

• one fasting blood sample to measure various hormones; fasting glucose:insulin ratio; pelvic ultrasound scan to determine ovarian morphology, follicular count and endometrial thickness

Part 1 of the research protocol will include obtaining the following:

* One urine & serum sample to be taken at the same time as their routine clinical blood samples.
* These samples will be anonymised before despatch to SPD. Part 2 of the study will involve treating patients with Vitamin D (if they are deficient) and/or myo-inositol supplement or metformin depending on their clinical need. The outcomes measured will be as above (blood sample to measure hormones) and an assessment of body fat distribution.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women with PCOS (Rotterdam criteria) attending the endocrine clinic, aged between 18-45 years

Exclusion Criteria:

* There is a clear exclusion criteria under the Rotterdam criteria; age <18 years or >45 years; oral contraceptive use within 3 months prior to recruitment, diabetes mellitus & pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female reproductive organs need to be present i.e. ovaries and uterus
Study Population: Women with polycystic ovary syndrome (PCOS)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-09-05 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Assay measurements of hormones in blood and urine samples i.e. testosterone, SHBG, FSH, LH, VD, AMH, fasting insulin & glucose. | 6 months
  Statistically significant differences in: levels of hormone/factors produced as measured in blood and urine samples sent to pathology lab; hormonal & metabolic responses/parameters after dietary/pharmaceutical intervention

SECONDARY OUTCOMES:
Measurement of BMI | 6 months
  BMI between different patient types

CONTACTS AND LOCATIONS:
Overall Officials: Suman Rice, PhD, Principal Investigator — St George's, University of London
Locations (1):
- St George's Hospital Trust, London, United Kingdom